CLINICAL TRIAL: NCT04698603
Title: A Phase 1/2 Study of GH001 in Patients With Treatment-Resistant Depression
Brief Title: Clinical Study of GH001 in Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GH Research Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GH001-TRD-102; 2018-004208-20 (EudraCT Number)
Record Dates: First submitted 2020-11-17; First posted 2021-01-07 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder; Depression
Keywords: Treatment; 5-MeO-DMT; 5-methoxy-dimethyltryptamine
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depression | interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Intervention Model Description: Phase 1 (Part A): Two dose levels of GH001 investigated in single doses. Phase 2 (Part B): GH001 investigated in an individualized dosing regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 (Part A): GH001 dose A (Experimental)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- Phase 1 (Part A): GH001 dose B (Experimental)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- Phase 2 (Part B): GH001 Individualized Dosing Regimen (Experimental)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine

INTERVENTIONS:
Drug: 5 Methoxy N,N Dimethyltryptamine — GH001 administered via inhalation
  Other Names: GH001; 5-MeO-DMT

SUMMARY:
The aim of the study is to investigate the safety of GH001 (containing 5-methoxy-dimethyltryptamine; 5-MeO-DMT), and to investigate its effects on severity of depressive symptoms, and its dose-related psychoactive effects in patients with Treatment-Resistant Depression (TRD).

The study is comprised of two open-label, single-arm study parts where Part A evaluates single doses of GH001 at two dose levels and Part B evaluates a specific individualized dosing regimen of GH001.

DETAILED DESCRIPTION:
Phase 1 (Part A):

The primary objective of this study is to assess the safety and tolerability of single doses of GH001 (containing 5-methoxy-dimethyltryptamine; 5-MeO-DMT) in patients with TRD.

The secondary objectives of the study are to assess the effects of single doses of GH001 on various measures of depression, and on dose-related psychoactive effects.

Phase 2 (Part B):

The primary objective of this study is to assess the effects of an individualized dosing regimen of GH001 on the severity of depression.

The secondary objectives of the study are to assess the safety and tolerability of an individualized dosing regimen of GH001 in patients with TRD and its effects on the severity of depression, other measures of depression, and on dose-related psychoactive effects.

Study design: Phase 1/2 study in two parts.

Intervention: In the Phase 1 (Part A), a single dose of GH001 will be administered per patient. Two different dose levels will be investigated with four patients at each dose level. In the Phase 2 (Part B), an individualized dosing regimen will be administered.

In both parts, GH001 will be administered via inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) in the range of 18.5 and 35.0 kg/m2 (inclusive);
* Meets the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) or recurrent MDD, without psychotic features confirmed by the Mini-International Neuropsychiatric Interview (MINI);
* Treatment-Resistant Depression as evaluated by the Antidepressant Treatment History Form - Short Form (ATHF-SF);
* Has outpatient status at screening and enrolment visits;

Exclusion Criteria:

* Has a current or prior diagnosis of a psychiatric comorbidity that renders the patient unsuitable for the study according to a study psychiatrist or registered psychologist;
* Has received any investigational medication within the last 1 month;
* Has a current medically significant condition (e.g., severe infection) or has a history of a medically significant condition (e.g., medical history of seizure, uncontrolled hypertension, uncontrolled diabetes, severe cardiovascular disease, hepatic or renal failure, etc.) that renders the patient unsuitable for the study according to the medical supervisor's judgment;
* Takes any medication or other substance that renders the patient unsuitable for the study according to the medical supervisor's judgment;
* Has a clinically significant abnormality in physical examination, vital signs, ECG, or clinical laboratory parameters, which renders the patient unsuitable for the study according to the medical supervisor's judgment;

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Phase 1: The safety and tolerability of GH001 as a combined measure of outcomes 5 to 13. | up to 7 days
  Phase 1: The primary endpoint is a binary variable (yes/no) reflecting a combined medical/clinical evaluation of the occurrence of Outcomes 5 to 13. The endpoint will be considered met for any dose level or regimen if the Study Safety Group (SSG) - through a qualitative medical/clinical evaluation - considers that dose level or regimen sufficiently safe and tolerable for potential further clinical development in a subsequent study.
Phase 2: The effects of GH001 on the severity of depression evaluated by the Montgomery-Asberg Depression Rating Scale (MADRS) | up to 7 days
  Phase 2: The assessment is done with the Montgomery-Asberg Depression Rating Scale (MADRS), a diagnostic questionnaire with ten items for measuring the severity of depressive episodes in patients with mood disorders. A higher MADRS score indicates more severe depression, and each item is scored from 0 to 6. The overall score ranges from 0 to 60.

SECONDARY OUTCOMES:
Phase 1: The effects of GH001 on the severity of depression evaluated by the Montgomery-Asberg Depression Rating Scale (MADRS) | up to 7 days
  Phase 1: The assessment is done with the Montgomery-Asberg Depression Rating Scale (MADRS), a diagnostic questionnaire with ten items for measuring the severity of depressive episodes in patients with mood disorders. A higher MADRS score indicates more severe depression, and each item is scored from 0 to 6. The overall score ranges from 0 to 60.
Phase 2: The safety and tolerability of GH001 as a combined measure of outcomes 5 to 13 | up to 7 days
  Phase 2: The secondary endpoint is a binary variable (yes/no) reflecting a combined medical/clinical evaluation of the occurrence of Outcomes 5 to 13. The endpoint will be considered met for any dose level or regimen if the Study Safety Group (SSG) - through a qualitative medical/clinical evaluation - considers that dose level or regimen sufficiently safe and tolerable for potential further clinical development in a subsequent study.

OTHER OUTCOMES:
Type and Frequency of Adverse Events | up to 7 days
  Adverse events reported in the study and coded by MedDRA.
Frequency of clinically significant changes from baseline in the safety laboratory analyses (biochemistry, hematology, urinalysis) | up to 7 days
  Safety laboratory analyses are analyses of blood samples (biochemistry, hematology) and urine samples (urinalysis). Changes are defined as any clinically significant change from baseline as determined by the medical supervisor at the site.
Frequency of clinically significant changes from baseline in Vital Signs | up to 7 days
  Vital signs include heart rate (beats per minute), blood pressure (mmHg), respiratory rate (breaths per minute), oxygen saturation (%), and temperature (degrees celsius). Changes are defined as any clinically significant change from baseline as determined by the medical supervisor at the site.
Frequency of clinically significant changes from baseline in Electrocardiogram (ECG) parameters | up to 3 hours after administration of GH001
  Clinically significant changes in ECG include any significant change in rate or rhythm as determined by the medical supervisor at the site.
Change from baseline in the Brief Psychiatric Rating Scale (BPRS) | up to 7 days
  Change from baseline in the Brief Psychiatric Rating Scale (BPRS). A scale to measure psychiatric symptoms. Each symptom is rated 1-7 and a total of 18 symptoms are scored. Combined score ranges from 18 to 126.
Change from baseline in the Clinician Administered Dissociative States Scale (CADSS) | up to 7 days
  Change from baseline in the Clinician Administered Dissociative States Scale (CADSS).
  The CADSS comprises 19 subjective items, ranging from 0 'not at all' to 4 'extremely. Summed together, these subscales form a total dissociative score. Combined score ranges from 0 to 76.
Change from baseline in the Columbia-Suicide Severity Rating Scale (C-SSRS) | up to 7 days
  Change from baseline in the Columbia-Suicide Severity Rating Scale (C-SSRS). A detailed questionnaire assessing both suicidal behaviour and suicidal ideation. No combined score is created.
Change from baseline in the Psychomotor Vigilance Test (PVT) | up to 7 days
  Change from baseline in the Psychomotor Vigilance Test (PVT). A computerized test assessing the reaction time in response to a visual stimulus. Outcome measures are Response Time and the number of attentional lapses (Response Time ≥ 500 msec).
Change from baseline in Digit Symbol Substitution Test (DSST) | up to 7 days
  Change from baseline in the Digit Symbol Substitution Test (DSST). A computerized test with the task is to match digits with symbols from encoding list. The number of digits correctly encoded within 3 minutes is the performance measure.

CONTACTS AND LOCATIONS:
Overall Officials: GH Research Clinical Team, Study Director — GH Research Ireland Limited
Locations (1):
- Clinical Trial Site, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reckweg JT, van Leeuwen CJ, Henquet C, van Amelsvoort T, Theunissen EL, Mason NL, Paci R, Terwey TH, Ramaekers JG. A phase 1/2 trial to assess safety and efficacy of a vaporized 5-methoxy-N,N-dimethyltryptamine formulation (GH001) in patients with treatment-resistant depression. Front Psychiatry. 2023 Jun 20;14:1133414. doi: 10.3389/fpsyt.2023.1133414. eCollection 2023. PMID 37409159